CLINICAL TRIAL: NCT04556981
Title: A Randomized, Placebo-controlled, Observer-blind, Phase 2 Study to Evaluate Safety and Immunogenicity of the Investigational M72/AS01E Mycobacterium Tuberculosis (Mtb) Vaccine in Virally Suppressed, Antiretroviral-treated Participants With Human Immunodeficiency Virus (HIV)
Brief Title: Safety and Immunogenicity of a Mycobacterium Tuberculosis Vaccine M72/AS01E in Participants With Well-controlled HIV
Acronym: MESA-TB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gates Medical Research Institute (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Gates MRI-TBV02-202; 221698/Z/20/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2020-09-10; First posted 2020-09-21 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Human Immunodeficiency Virus
Keywords: Mycobacterium tuberculosis; M72/AS01E Vaccine; Antiretroviral therapy; Mtb; HIV; TB vaccine
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- M72/AS01E vaccine (Experimental)
  Interventions: Biological: M72/AS01E Mycobacterium tuberculosis vaccine
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: M72/AS01E Mycobacterium tuberculosis vaccine — Participants will receive an intramuscular dose of M72 (10 micrograms of recombinant fusion protein) reconstituted with AS01E (an adjuvant system), on Day 1 and Day 29
  Arms: M72/AS01E vaccine
Biological: Placebo — Participants will receive an intramuscular dose of saline (0.9% NaCl), on Day 1 and Day 29
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of M72/AS01E vaccination in virally suppressed, antiretroviral-treated participants with human immunodeficiency virus infection (HIV).

ELIGIBILITY:
Inclusion Criteria:

* Participant with documented human immunodeficiency virus (HIV) infection who fulfill all of the following:

  * Has reactive anti-HIV antibody at screening
  * On antiretroviral therapy (ART) for at least 3 consecutive months at screening
  * Has documented HIV RNA <200 copies/mL at screening
  * Participants with CD4+ cell counts ≥200 cells/μL at screening
* Participants have had tuberculosis (TB) preventive therapy (TPT) in the past and are not receiving TPT at the time of screening, according to the judgment of the investigators
* Participants who are healthy as determined by medical evaluation including medical history, physical examination and laboratory tests
* Capable of giving signed informed consent and informed assent (if appropriate), which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) or informed assent form, and in the protocol.
* Female participants of childbearing potential must agree not to become pregnant from the time of study enrollment for one year after study intervention. Women physically capable of pregnancy, sexually active and having no history of hysterectomy or tubal ligation or menopause must agree to use an effective method of avoiding pregnancy during this period.
* Participants who agree to stay in contact with the study site for the duration of the study, provide updated contact information as necessary, and have no current plans to relocate from the study area for the duration of the study.

Exclusion Criteria:

* Acute illness or fever ≥99.5°F (or ≥37.5˚C) on Day 1
* History of active TB disease
* Evidence of active TB disease with any of the following:

  * Have symptoms or signs of TB disease
  * Have a positive sputum Xpert MTB/RIF assay (only in participants with sputum sample at screening)
  * Are on treatment for active TB disease
* Evidence and/or history of clinically significant medical conditions (other than HIV infection) as judged by the investigator, including malignancies
* Any current medical, psychiatric, occupational, or substance abuse problems that, in the opinion of the investigator, will make it unlikely that the participant will comply with the protocol
* Any medications or other therapies that may impact the immune system such as immune globulin, interferon, immunomodulators, cytotoxic drugs or other drugs known to be frequently associated with major organ toxicity as determined by the investigator, within 90 days prior to Day 1
* Immunosuppressive agents including systemic steroids - prior corticosteroid therapy within 90 days prior to Day 1 (permitted: 5 mg/day prednisone equivalent, inhaled, topical, and intra-articular corticosteroids)
* Receipt or donation of blood or blood products within 90 days prior to Day 1 or planned receipt or donation during the study period
* Participation in an interventional clinical trial and/or receipt of any investigational drug within 180 days prior to signing informed consent or assent
* Receipt of any vaccine in the period starting 7 days before, and ending 7 days after, each dose of the study vaccine
* History of previous administration of experimental Mycobacterium tuberculosis vaccine
* Safety laboratory values outside of normal range, for age and sex that are suggestive of a disease state (Grade 1 abnormalities, as per Division of AIDS [DAIDS] toxicity table version 2.1, will not lead to exclusion if the investigator considers them not clinically significant.)
* Urinalysis abnormality greater than Grade 1 on the Toxicity Scale (with the exception of hematuria in a menstruating female), or urinalysis abnormality judged clinically significant by the investigator
* Current hepatitis B and/or hepatitis C infection
* Indeterminate QFT result
* History of allergy or hypersensitivity to the study drug, excipients or related substances
* Shared residence with an individual who is receiving TB treatment or with someone who is known to have incompletely treated TB, e.g., Xpert MTB/RIF assay-positive, polymerase chain reaction (PCR)-positive, culture-positive, smear-positive TB, or clinically diagnosed unconfirmed TB
* Female participants with any one of the following conditions: currently pregnant or lactating/nursing; having positive serum pregnancy test during the screening window, planning a pregnancy within 1 year after first dose of study product
* Individuals who are acting as study personnel or immediate family members (brother, sister, child, parent) or the spouse/partner of study personnel.
* Child in Care

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 402 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gates MRI, Study Director — Gates Medical Research Institute
Locations (6):
- South Africa (6):
  - Wits RHI, Johannesburg, Gauteng
  - Ekhaya VAC, Cape Town, Khayelitsha
  - CAPRISA, Durban, KwaZulu-Natal
  - The Aurum Institute, Klerksdorp, North West
  - Desmond Tutu HIV Foundation, Cape Town, Western Cape
  - SATVI, Worcester, Western Cape

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Dagnew AF, Han LL, Naidoo K, Fairlie L, Innes JC, Middelkoop K, Tameris M, Wilkinson RJ, Ananworanich J, Bower D, Schlehuber L, Frahm N, Cinar A, Dunne M, Schmidt AC. Safety and immunogenicity of investigational tuberculosis vaccine M72/AS01E-4 in people living with HIV in South Africa: an observer-blinded, randomised, controlled, phase 2 trial. Lancet HIV. 2025 Aug;12(8):e546-e555. doi: 10.1016/S2352-3018(25)00124-9. Epub 2025 Jul 1. PMID 40614747

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in South Africa.
Pre-assignment Details: This was a randomized, placebo-controlled, observer-blind, phase 2 study to evaluate safety and immunogenicity of the investigational M72/AS01E Mycobacterium tuberculosis (Mtb) vaccine in virally suppressed, antiretroviral-treated participants with human immunodeficiency virus (HIV).
Groups:
- M72/AS01E: Participants were randomized to receive an intramuscular dose of M72/AS01E: M72 (10 micrograms of recombinant fusion protein) reconstituted with AS01E (an adjuvant system), on Day 1 and Day 29
- Placebo: Participants were randomized to receive an intramuscular dose of placebo (saline [0.9% sodium chloride {NaCl}]), on Day 1 and Day 29
Period: Overall Study
Arm/Group | M72/AS01E | Placebo
Started | 202 | 200
Completed | 195 | 181
Not Completed | 7 | 19
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 2 | 11
Not completed — Moved from the study area | 1 | 4
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: included all participants randomly assigned to study intervention and who received at least one dose of study intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | M72/AS01E | Placebo | Total
Number analyzed (Participants) | 201 | 200 | 401
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.4 (4.17) | 29.6 (4.47) | 29.5 (4.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 175 | 176 | 351
  Male | 26 | 24 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 201 | 200 | 401
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 196 | 196 | 392
  Southern African Coloured | 5 | 4 | 9
QuantiFERON®-TB Gold Plus assay status [Count of Participants; unit: Participants]
  Positive | 93 | 100 | 193
  Negative | 108 | 100 | 208
Cluster of differentiation 4 (CD4+) [Number; unit: 10^6 cells/liter (L)]
  <200*10^6 cells/L | 0 | 0 | 0
  200-349*10^6 cells/L | 7 | 5 | 12
  350-499*10^6 cells/L | 20 | 24 | 44
  >=500*10^6 cells/L | 174 | 171 | 345
Human immunodeficiency virus (HIV) ribonucleic acid (RNA) viral load [Number; unit: copies per mL]
  Not Detected | 162 | 162 | 324
  <=200 copies per mL | 36 | 35 | 71
  >200 copies per mL | 3 | 3 | 6
Weight [Mean (Standard Deviation); unit: Kilograms] | 73.4 (19.93) | 74.3 (18.81) | 73.8 (19.36)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Adverse Events (AEs) Through 7 Days Post Dose 1 of Study Intervention
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An AE does not necessarily have a causal relationship with the intervention. Solicited AEs were defined events that participants were specifically asked about and which were noted by participants in the diary card. Solicited local AEs included pain, redness and swelling and general body symptoms such as fever, headache, fatigue, gastrointestinal symptoms, and myalgia.
Time Frame: Day 1 through Day 7 (after first vaccination)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | M72/AS01E | Placebo
Number analyzed (Participants) | 201 | 200
Participants
  Any injection site symptom | 155 | 49
  Any general body symptom | 132 | 109

2. Primary Outcome: Number of Participants With Solicited AEs Through 7 Days Post Dose 2 of Study Intervention
Description: as for outcome 1
Time Frame: Day 29 through Day 35 (after second vaccination)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | M72/AS01E | Placebo
Number analyzed (Participants) | 201 | 200
Participants
  Any injection site symptom | 147 | 29
  Any general body symptom | 134 | 83

3. Primary Outcome: Number of Participants With Unsolicited AEs Through 28 Days Post Dose 1 of Study Intervention
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An AE does not necessarily have a causal relationship with the intervention. Unsolicited AEs were all AEs for which the participant was not specifically questioned in the participant diary card. Number of Participants With Unsolicited AEs Through 28 Days after first vaccination has been presented.
Time Frame: Day 1 through Day 28
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | M72/AS01E | Placebo
Number analyzed (Participants) | 201 | 200
Participants | 67 | 67

4. Primary Outcome: Number of Participants With Unsolicited AEs Through 28 Days Post Dose 2 of Study Intervention
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An AE does not necessarily have a causal relationship with the intervention. Unsolicited AEs were all AEs for which the participant was not specifically questioned in the participant diary card. Number of Participants With Unsolicited AEs Through 28 Days after second vaccination has been presented.
Time Frame: Day 29 through Day 57
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | M72/AS01E | Placebo
Number analyzed (Participants) | 185 | 188
Participants | 53 | 41

5. Primary Outcome: Number of Participants Reporting Serious AEs (SAEs)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment. Number of Participants reporting SAEs has been presented.
Time Frame: Up to Day 390
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | M72/AS01E | Placebo
Number analyzed (Participants) | 201 | 200
Participants | 4 | 5

6. Secondary Outcome: Number of Participants With Potential Immune-mediated Diseases (pIMDs)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. pIMDs are a subset of AEs that included autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology. Number of Participants With Potential Immune-mediated Diseases (pIMDs) has been presented
Time Frame: Up to Day 390
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | M72/AS01E | Placebo
Number analyzed (Participants) | 201 | 200
Participants | 0 | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Hematology Assessments of Grade 3 or Above After Baseline
Description: Blood samples were collected for the assessment of hemoglobin, leukocytes and platelets. Baseline was defined as last non-missing assessment prior to first vaccination. Laboratory grades were evaluated using the Common Terminology Criteria for AEs (CTCAE version (v)5.0) with grading as: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life-threatening or disabling. Number of Participants With Clinically Significant hematology assessments of Grade 3 and Grade 4 has been presented.
Time Frame: Up to Day 390
Population: Safety Population. Only those participants with data available at the specified data points were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | M72/AS01E | Placebo
Number analyzed (Participants) | 197 | 191
Participants
  Hemoglobin: Grade 3 | 0 | 0
  Hemoglobin: Grade 4 | 0 | 0
  Leukocytes: Grade 3 | 0 | 0
  Leukocytes: Grade 4 | 0 | 0
  Platelets: Grade 3 | 0 | 0
  Platelets: Grade 4 | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Chemistry Assessments of Grade 3 or Above After Baseline
Description: Blood samples were collected for the assessment of Alanine Aminotransferase, Aspartate Aminotransferase and total bilirubin. Baseline was defined as last non-missing assessment prior to first vaccination. Laboratory grades were evaluated using the CTCAE v5.0 with grading as: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Life-threatening or disabling. Number of Participants With Clinically Significant chemistry assessments of Grade 3 and Grade 4 has been presented.
Time Frame: Up to Day 390
Population: Safety Population. Only those participants with data available at the specified data points were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | M72/AS01E | Placebo
Number analyzed (Participants) | 197 | 191
Participants
  Alanine Aminotransferase: Grade 3 | 0 | 1
  Alanine Aminotransferase: Grade 4 | 0 | 0
  Aspartate Aminotransferase: Grade 3 | 0 | 1
  Aspartate Aminotransferase: Grade 4 | 0 | 0
  Total bilirubin: Grade 3 | 0 | 0
  Total bilirubin: Grade 4 | 0 | 0

9. Secondary Outcome: M72-specific Antibody Titers
Description: Blood samples for immunogenicity evaluation of M72-specific IgG antibody in serum were collected. On Day 1 and Day 29 visits, samples were collected prior to study intervention administration. Humoral M72-specific IgG antibodies were measured by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 1, Day 29, Day 57, Day 210 and Day 390
Population: Per-Protocol (PP) Population: included all participants randomly assigned to study intervention, who received the study interventions as planned and did not substantially deviate from the protocol procedures. Only those participants with data available at the specified data points were analyzed
Measure: Geometric Mean (95% Confidence Interval); unit: Equivalent units per mL (EU/mL)
Arm/Group | M72/AS01E | Placebo
Number analyzed (Participants) | 143 | 130
Equivalent units per mL (EU/mL)
  Day 1 | 2.72 [2.69 to 2.76] | 2.77 [2.69 to 2.85]
  Day 29 | 13.28 [10.99 to 16.04] | 2.77 [2.69 to 2.86]
  Day 57 | 479.70 [421.79 to 545.56] | 2.77 [2.69 to 2.86]
  Day 210 | 52.23 [44.83 to 60.86] | 2.77 [2.70 to 2.85]
  Day 390: number analyzed (Participants) | 142 | 129
  Day 390 | 32.43 [27.94 to 37.65] | 2.77 [2.69 to 2.85]

10. Secondary Outcome: Number of M72 Specific CD4+ and CD8+ T Cell Responders Based on Cytokine Response
Description: Blood samples were analyzed for M72-specific CD4+ and CD8+ T-cell responses based on IFN-gamma and/or IL-2 expression. The CD4+ and CD8+ categories for each timepoint are mutually exclusive.
Time Frame: Day 57 and Day 390
Population: Per-Protocol for Cellular Immunogenicity Population comprises all participants in PP population randomly selected to have immunogenicity assays performed. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | M72/AS01E | Placebo
Number analyzed (Participants) | 96 | 32
Participants
  CD4+ Responders on Day 57: number analyzed (Participants) | 96 | 31
  CD4+ Responders on Day 57 | 92 | 6
  CD4+ non-responders on Day 57: number analyzed (Participants) | 96 | 31
  CD4+ non-responders on Day 57 | 4 | 25
  CD4+ Responders on Day 390 | 85 | 8
  CD4+ non-responders on Day 390 | 11 | 24
  CD8+ Responders on Day 57: number analyzed (Participants) | 96 | 31
  CD8+ Responders on Day 57 | 14 | 3
  CD8+ non-responders on Day 57: number analyzed (Participants) | 96 | 31
  CD8+ non-responders on Day 57 | 82 | 28
  CD8+ Responders on Day 390 | 10 | 3
  CD8+ non-Responders on Day 390 | 86 | 29

11. Secondary Outcome: Percentage of M72-specific CD4+ T Cells and CD8+ T Cells Exhibiting Cytokine Response With Background Subtracted
Description: Blood samples were analyzed for M72-specific CD4+ and CD8+ T-cells exhibiting cytokine response (IFN-gamma and/or IL-2) with background subtracted. Baseline is defined as the last non-missing assessment (scheduled or unscheduled) prior to the first study vaccination.
Time Frame: At Baseline, Day 57, and Day 390
Population: Per-Protocol for Cellular Immunogenicity Population comprises all participants in Per-Protocol population randomly selected to have immunogenicity assays performed. Only those participants with data available at specified timepoints has been presented.
Measure: Mean (Standard Deviation); unit: Percentage of cells
Arm/Group | M72/AS01E | Placebo
Number analyzed (Participants) | 96 | 32
Percentage of cells
  CD4+ at Baseline | 0.062 (0.506) | 0.067 (0.167)
  CD4+ at Day 57: number analyzed (Participants) | 96 | 31
  CD4+ at Day 57 | 0.534 (0.556) | 0.014 (0.096)
  CD4+ at Day 390 | 0.339 (0.375) | 0.047 (0.169)
  CD8+ at Baseline | 0.071 (0.248) | 0.092 (0.353)
  CD8+ at Day 57: number analyzed (Participants) | 96 | 31
  CD8+ at Day 57 | 0.092 (0.272) | -0.007 (0.042)
  CD8+ at Day 390 | 0.090 (0.328) | 0.058 (0.371)

ADVERSE EVENTS:
Time Frame: Solicited AEs (comprising of injection site pain, redness, swelling, headache, fatigue, myalgia, gastrointestinal symptoms, and pyrexia) were recorded on diary cards (systematic assessment) for 7 days after each dose. Solicited events ongoing at Day 7 were collected as unsolicited AEs. Unsolicited AEs were collected through 28 days after each dose, and SAEs (non-systematic assessments) were collected from dosing at Day 1 through Day 390 (end of study).
Description: An AE was classified as solicited if it was proactively recorded through a structured assessment (e.g., diary card) through 7 days post vaccination. A participant who had an event ongoing at Day 7 would have the event counted as both a solicited AE and an unsolicited AE.
Arm/Group | M72/AS01E | Placebo
All-Cause Mortality (participants affected / at risk) | 0/201 | 1/200
Serious Adverse Events (participants affected / at risk) | 4/201 | 5/200
Other Adverse Events (participants affected / at risk) | 191/201 | 158/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | M72/AS01E (N=201) | Placebo (N=200)
COVID-19 (Infections and infestations) | 1 | 1
Anal abscess (Infections and infestations) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 1
Physical assault (Social circumstances) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | M72/AS01E (N=201) | Placebo (N=200)
Conjunctivitis allergic (Eye disorders) | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 2
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1
Toothache (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2
Injection site erythema (General disorders) | 12 | 1
Influenza like illness (General disorders) | 6 | 3
Injection site pruritus (General disorders) | 5 | 1
Injection site swelling (General disorders) | 18 | 0
Pyrexia (General disorders) | 3 | 4
Injection site pain (General disorders) | 11 | 0
Fatigue (General disorders) | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 5
Influenza (Infections and infestations) | 4 | 6
Tonsillitis (Infections and infestations) | 3 | 0
Rhinitis (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 4
Conjunctivitis (Infections and infestations) | 0 | 2
Alanine aminotransferase increased (Investigations) | 4 | 5
Aspartate aminotransferase increased (Investigations) | 3 | 6
Blood pressure increased (Investigations) | 3 | 1
Haemoglobin decreased (Investigations) | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Headache (Nervous system disorders) | 23 | 30
Dizziness (Nervous system disorders) | 8 | 9
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 2 | 4
Menorrhagia (Reproductive system and breast disorders) | 0 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 4 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Injection site pain (General disorders) | 167 | 50
Injection site erythema (General disorders) | 67 | 19
Injection site swelling (General disorders) | 83 | 17
Headache (Nervous system disorders) | 132 | 78
Fatigue (General disorders) | 119 | 74
Gastrointestinal symptoms (Gastrointestinal disorders) | 56 | 38
Myalgia (Musculoskeletal and connective tissue disorders) | 96 | 45
Pyrexia (General disorders) | 87 | 44
Nausea (Gastrointestinal disorders) | 1 | 2
Chest pain (General disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT04556981/Prot_002.pdf
  • Statistical Analysis Plan (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/81/NCT04556981/SAP_003.pdf